CLINICAL TRIAL: NCT02233075
Title: A Study of the Safety and Efficacy of Combination Treatment With REP 2139-Ca and Pegasys™ in Patients With Hepatitis B / Hepatitis D Co-infection
Brief Title: REP 2139-Ca / Pegasys™ Combination Therapy in Hepatitis B / Hepatitis D Co-infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Replicor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REP 301
Record Dates: First submitted 2014-09-01; First posted 2014-09-08 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-02

CONDITIONS: Chronic HBV Infection (HBeAg Negative)
MeSH Terms: interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- REP 2139-Ca + Pegasys (TM) (Experimental): REP 2139-Ca 500 mg QW for 15 weeks followed by REP 2139-Ca 250mg QW + Pegasys(TM) 180ug QW for 15 weeks followed by Pegasys(TM) 180ug QW for 33 weeks.
  Interventions: Drug: REP 2139-Ca + Pegasys (TM)

INTERVENTIONS:
Drug: REP 2139-Ca + Pegasys (TM) — 15 weeks of REP 2139-Ca (500mg QW IV) followed by: 15 weeks of REP 2139-Ca (250mg QW IV) + Pegasys(TM) (180 ug QW SC) followed by: 33 weeks of Pegasys(TM) (180 ug QW SC)
  Other Names: Pegasys(TM) = pegylated interferon alpha-2a

SUMMARY:
REP 2139-Ca is nucleic acid polymer. Nucleic acid polymers have been previously shown to clear serum hepatitis B virus surface antigen (HBsAg) both preclinically (in duck HBV infected ducks) and in human patients and to act synergistically with immunotherapeutic agents such as pegylated interferon-alpha 2a or thymosin alpha-1 to restore host immunological control of HBV infection.

HBsAg is an essential component of the hepatitis D virus (HDV), therefore the direct action of REP 2139-Ca in removing serum HBsAg and its synergistic effect with pegylated interferon-alpha 2a is expected to have a significant antiviral effect against HDV infection.

This study will examine the safety and efficacy of REP 2139-Ca therapy when used in combination with pegylated interferon alpha-2a in patients with HBV / HDV co-infection.

The primary hypothesis to be tested is that this combined dosing regimen is safe and well tolerated in patients with HBV / HDV co-infection which will be assessed by examining the number of patients with adverse events (including reported symptoms and laboratory abnormalities).

The secondary hypothesis to be tested is that this combined dosing regimen will have an antiviral effect against HBV / HDV co-infection in these patients which will be assessed by examining the following outcomes:

1. The number of patients with reductions in serum HBsAg.
2. The number of patients with reductions in serum HDAg and HDV RNA
3. The number of patients that experience a sustained antiviral response after treatment is stopped (reductions in serum HBV DNA and HDV RNA).

The secondary hypothesis to be tested is that this combination approach can have an effective

DETAILED DESCRIPTION:
Nucleic acid polymers (NAPs) utilize the sequence independent properties of phosphorothioated oligonucleotides to target apolipoprotein interactions involved in the formation of HBV subviral particles (SVPs) which are comprised mainly of the hepatitis B surface antigen protein (HBsAg). The effect of NAPs is to block the formation of SVPs inside infected hepatocytes which prevents their secretion. As SVPs account for > 99.99% of HBsAg in the blood, NAPs are an effective approach for clearing HBsAg from the serum of HBV infected patient.

Previous clinical trials have demonstrated that treatment with the NAP REP 2139 results in the rapid and effective clearance of HBsAg from the blood. This HBsAg removal has the immediate effect of unmasking the underlying, pre-existing anti-HBsAg (anti-HBs) response, allowing clearance of HBV virus from the blood.

HBsAg has important immunosuppressive effects in HBV infection which have been shown to block both adaptive and innate immune processes. Removal of HBsAg from the blood of patients removes this immunosuppressive effect.

Thus, an important additional effect of removal of HBsAg from the blood is to greatly enhance the effect of immunotherapeutic agents like pegylated interferon alpha-2a or thymosin alpha-1 to stimulate recovery of complete immune control of HBV infection.

HDV superinfection can only occur in patients with HBV infection because HDV requires the HBsAg protein for its assembly. Therefore, it is expected that the removal of serum HBsAg (from HBV SVPs) and unmasking of the anticipated, pre-existing anti-HBsAg response by REP 2139 will result in the clearance of HBV and HDV from the blood. Furthermore, the enhanced effect of immunotherapy in the absence of serum HBsAg has the potential to provide a durable control of both HBV and HDV infection that will persist after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years
* HBsAg > 1000 IU / ml
* HDAg+
* HDV RNA +
* No detectable antibodies to HIV, HCV or CMV.
* Non cirrhotic
* Willingness to utilize adequate contraception while being treated with REP 213-Ca and for 6 months following the end of treatment
* Adequate venous access allowing weekly intravenous therapies and blood tests
* Body Mass Index (BMI) ≥ 18 kg/m2 and ≤ 25 kg/m2

Exclusion Criteria:

* Evidence of cardiovascular disease
* Evidence of autoimmune hepatitis
* Presence of Wilson's disease
* Presence of severe NAFLD
* Evidence of any other co-existent liver disease
* ANA (anti-nuclear antibody) positive
* Fibroscan and Fibromax showing evidence of advanced cirrhosis.
* Any history of ascites, hepatic encephalopathy or variceal hemorrhage
* Body weight > 100 kg
* Platelet count < 90,000, PMN count < 1,500 or HCT < 33%
* Evidence of significant heavy metal load in whole blood.
* AFP > 100 ng/ml or the presence of a hepatic mass suggestive of HCC
* Bilirubin above the normal range
* ALT > 5x ULN
* Creatinine > 1.5 mg/dl
* Serum albumin < 35 mg/ml
* The presence of diabetes (whether controlled or uncontrolled)
* Another serious medical disorder
* A serious psychiatric disorder
* Evidence of hypertension
* A history of alcohol abuse within the last year
* The use of illicit drugs within the past two years
* Inability to provide informed consent
* Inability or unwillingness to provide weekly blood samples
* Poor venous access making IV infusion too difficult
* Patient not willing to come every week to receive therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing a treatment-related adverse event. | Every week for 63 weeks.
  Will examine the hypothesis that combined REP 2139-Ca / Pegasys(TM) treatment is safe and well tolerated in patients with HBV / HDV co-infection

SECONDARY OUTCOMES:
Number of patients with reduction of serum HBsAg. | Every two weeks for 63 weeks (treatment duration) + 24 weeks (follow-up)
  Will examine the hypothesis that combination treatment with REP 2139-Ca / Pegasys(TM) will have an antiviral effect in patients with HBV / HDV co-infection.
Number of patients with reduced serum HDV antigen / HDV RNA | Every two weeks for 63 weeks (treatment duration) + 24 weeks followup
  Will examine the hypothesis that combination treatment with REP 2139-Ca / Pegasys(TM) will have an antiviral effect in patients with HBV / HDV co-infection.
Number of patients with controlled HBV / HDV infection following treatment | 24 weeks follow up (after completion of 63 weeks of treatment)
  Will examine the hypothesis that combination treatment with REP 2139-Ca / Pegasys(TM) will have an antiviral effect in patients with HBV / HDV co-infection.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Pantea, MD, Principal Investigator — Infectious Diseases Department, State University of Medicine and Pharmacy
Locations (1):
- Infectious Clinical Hospital ( n.a. Toma Ciorba), Chisinau, Moldova

REFERENCES:
- [Background] Noordeen F, Vaillant A, Jilbert AR. Nucleic acid polymers inhibit duck hepatitis B virus infection in vitro. Antimicrob Agents Chemother. 2013 Nov;57(11):5291-8. doi: 10.1128/AAC.01003-13. Epub 2013 Aug 12. PMID 23939902
- [Background] Noordeen F, Vaillant A, Jilbert AR. Nucleic acid polymers prevent the establishment of duck hepatitis B virus infection in vivo. Antimicrob Agents Chemother. 2013 Nov;57(11):5299-306. doi: 10.1128/AAC.01005-13. Epub 2013 Aug 12. PMID 23939904
- [Derived] Bazinet M, Pantea V, Cebotarescu V, Cojuhari L, Jimbei P, Anderson M, Gersch J, Holzmayer V, Elsner C, Krawczyk A, Kuhns MC, Cloherty G, Dittmer U, Vaillant A. Persistent Control of Hepatitis B Virus and Hepatitis Delta Virus Infection Following REP 2139-Ca and Pegylated Interferon Therapy in Chronic Hepatitis B Virus/Hepatitis Delta Virus Coinfection. Hepatol Commun. 2020 Nov 13;5(2):189-202. doi: 10.1002/hep4.1633. eCollection 2021 Feb. PMID 33553968
- [Derived] Bazinet M, Pantea V, Cebotarescu V, Cojuhari L, Jimbei P, Albrecht J, Schmid P, Le Gal F, Gordien E, Krawczyk A, Mijocevic H, Karimzadeh H, Roggendorf M, Vaillant A. Safety and efficacy of REP 2139 and pegylated interferon alfa-2a for treatment-naive patients with chronic hepatitis B virus and hepatitis D virus co-infection (REP 301 and REP 301-LTF): a non-randomised, open-label, phase 2 trial. Lancet Gastroenterol Hepatol. 2017 Dec;2(12):877-889. doi: 10.1016/S2468-1253(17)30288-1. Epub 2017 Sep 28. PMID 28964701